CLINICAL TRIAL: NCT04279158
Title: Attention Modulation of Local and Global Inhibition Mechanisms
Acronym: MILGattention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0728; 2019-A03055-52 (Other: ID-RCB)
Record Dates: First submitted 2020-02-11; First posted 2020-02-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Optical Phenomena
Keywords: attention-deficit hyperactivity disorder (ADHD); Attention Deficit Disorder with Hyperactivity; attention; inhibition; Healthy Volunteers; Perceptual Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Inhibition, Psychological; Perceptual Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients with optic ataxia (OA) (Experimental)
  Interventions: Behavioral: experience 1 "The negative priming task"; Behavioral: experience 2 "Stop signal task"; Behavioral: experience 3 "Anti-saccades"
- patients with hemispatial neglect (Experimental)
  Interventions: Behavioral: experience 1 "The negative priming task"; Behavioral: experience 2 "Stop signal task"; Behavioral: experience 3 "Anti-saccades"
- patients with attention-deficit hyperactivity disorder (Experimental)
  Interventions: Behavioral: experience 1 "The negative priming task"; Behavioral: experience 2 "Stop signal task"; Behavioral: experience 3 "Anti-saccades"
- Healthy volunteers (Active Comparator)
  Interventions: Behavioral: experience 1 "The negative priming task"; Behavioral: experience 2 "Stop signal task"; Behavioral: experience 3 "Anti-saccades"

INTERVENTIONS:
Behavioral: experience 1 "The negative priming task" — The targets are presented to the subject on a computer screen. The subject must make an eye or hand movement toward the target and ignore the distracters.
Behavioral: experience 2 "Stop signal task" — The targets are presented to the subject on a computer screen. The subject must make an eye movement towards this target. Sometimes a stop signal will appear and the subject will have to avoid to look at the target
Behavioral: experience 3 "Anti-saccades" — The targets are presented to the subject on a computer screen. The subject must make an eye movement toward this target. Sometimes an instruction will ask the subject to look at the opposite of the target

SUMMARY:
Human behavior is both flexible and adapted to the environmental context through inhibition capabilities; the investigator control the subject's behavior by repressing inappropriate responses and selecting, among several possibilities, those that are appropriate. These mechanisms are not independent of attentional control. Attention acts as a selection filter for the investigator's behavior. This leads us to hypothesize that attention modulates the mechanisms of inhibition. Nevertheless, the different brain structures involved, as well as mechanisms underlying the interaction between inhibition and attention remain largely unknown.

Previous research has suggested that inhibition requires selective attention and, conversely, attentional mechanisms would result in the "deselection", or inhibition, of objects in space or irrelevant actions. Reconciling the literature on attention with the one on inhibition appears fundamental for the understanding of the instance to which the mechanisms of inhibition and the cognitive processes interact. Therefore, the goal of this research project will be to investigate how inhibition mechanisms are implemented in the brain and, in more detail, what determines the type of resulting inhibitory control: spatially localized or global. The investigator will test 3 different patient groups (optic ataxia, hemispatial neglect and attention-deficit hyperactivity disorder) compared to control.

In conclusion, this research project will aim to develop a theoretical model of the interaction between attentional control and inhibition mechanisms in order to improve diagnostic and rehabilitation tools in the future.

ELIGIBILITY:
All patients and healthy subjects:

Inclusion Criteria:

* male and female, age from 18 to 75 years included
* normal vision or corrected vision
* covered by social security
* signed written informed consent

Exclusion Criteria:

* unable to comply with requirements of the study (neurological, psychiatric, sensory or motor troubles)
* adults under legal protection

Patient with hemispatial neglect:

Inclusion Criteria:

* After a stroke (> 1 month ago), presence of a neurological impairment documented by brain imaging (standard of care) and by clinical symptoms.
* The diagnosis will be dissociated from hemianopia by perimetry. The hemispatial neglect consists of a lack of perception and responsiveness concerning the controlesional visual hemifield.

Patient with optic ataxia:

* After a stroke (> 1 month ago), presence of neurological injury in parietal cortex only, supported by a standard of care cerebral MRI
* Present optic ataxia symptoms (The OA consists of pointing errors with the hand contralateral to the lesion (hand effect) and / or to visual targets presented in the field contralateral to the lesion (field effect)).

Patient (adult and children) with attention-deficit hyperactivity disorder:

* present a diagnosis of ADHD subtype inattention or impulse / hyperactivity as established by a neuropsychologist.
* Children will be between 8 and 18 years old
* Adults will be between 18 and 75 years old.
* Participants will not report any comorbid learning disabilities to ADHD.

For minors:

- Having obtained the written consent of the legal representative(s)

Healthy subjects

Inclusion Criteria:

- no known neurological injury

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2031-11-26 (Estimated); Study Completion 2031-11-26 (Estimated)

PRIMARY OUTCOMES:
error rate | at the end of the simulation passage, an average of 3 years
  The investigator calculate the number of right and wrong answers (a correct answer is a saccade carried out when it is necessary and by reaching the target; a false answer is a saccade made at the wrong time and / or not reaching the target) to obtain the error rate.

SECONDARY OUTCOMES:
reaction time | at the end of the simulation passage, an average of 3 years
  The investigator measure the time it takes for the subject to respond (perform the eye saccade)

CONTACTS AND LOCATIONS:
Overall Officials: Laure PISELLA, Principal Investigator — Centre de recherche de Neurosciences de Lyon (CRNL)
Locations (1):
- Centre de Recherche en Neuroscience de Lyon, Bron, France